CLINICAL TRIAL: NCT07212816
Title: Detection of Atrial Fibrillation Through Voice Signal Processing
Status: Not yet recruiting | Type: Observational
Sponsor: Vital Audio Inc (Other)
Collaborators: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Sonometrik-AFIB-01
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation (AF); Atrial Flutter
Keywords: Cardioversion; Irregular Heart Rhythm; Arrhythmia; Atrial Fibrillation; Afib; Artificial Intelligence (AI) in Cardiology; Digital Biomarkers; Voice Biomarkers; Voice Signal Processing; Voice based monitoring
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Atrial Fibrillation Patients Undergoing Cardioversion: Investigational, software-only device that acquires short voice samples during automated phone calls and analyzes cardiopulmonary signals to estimate heart rate (HR), heart-rate variability (HRV), and rhythm status (regular vs irregular). In this study, three calls are initiated via the Vital Audio web platform (pre-, post-cardioversion, and 1-month follow-up). Results are available only to study staff and are compared with ECG obtained at the same time points. The device is used for data collection/assessment only and does not guide clinical care. IDE: G230147.
  Interventions: Device: Sauti

INTERVENTIONS:
Device: Sauti — Investigational, software-only device that acquires short voice samples during automated phone calls and analyzes cardiopulmonary signals to estimate heart rate (HR), heart-rate variability (HRV), and rhythm status (regular vs irregular). In this study, three calls are initiated via the Vital Audio web platform (pre-, post-cardioversion, and 1-month follow-up). Results are available only to study staff and are compared with ECG obtained at the same time points. The device is used for data collection/assessment only and does not guide clinical care. IDE: G230147.

SUMMARY:
This study is testing a new technology that listens to a person's voice during short phone calls to help identify heart rhythm problems. The goal is to see if voice signal analysis can tell the difference between a normal rhythm (sinus rhythm) and an irregular rhythm (atrial fibrillation).

We are enrolling adults scheduled for a standard heart procedure called cardioversion, which is used to reset the heart to a normal rhythm. Each participant will provide voice recordings through three short phone calls: before cardioversion, just after the procedure, and at a follow-up visit. Results will be compared with standard heart rhythm tests (electrocardiograms or ECGs).

This research may lead to a simple, low-cost way to monitor heart rhythms remotely without requiring special devices.

DETAILED DESCRIPTION:
This is a prospective, single-center cohort study of 40 patients undergoing cardioversion for atrial fibrillation at the Minneapolis Heart Institute Foundation. The study is designed to evaluate whether Vital Audio's investigational vocal biomarker software can reliably distinguish between regular (sinus) and irregular (atrial fibrillation) heart rhythms.

Participants will serve as their own controls. They will complete three structured voice recordings: pre-cardioversion, immediately after cardioversion, and at a follow-up visit (1 week to 1 month later). At each time point, ECG data will be collected as the reference standard. Voice samples will be captured through automated phone calls initiated via the Vital Audio platform, with each call lasting about one minute.

The software analyzes short vowel sounds in real time to extract heart rate, heart rate variability, and rhythm classification (regular vs. irregular). Data are stored securely, and results are available only to study staff. Patients and their providers will not receive study results directly.

The study is minimal risk, with no cost to participants. Compensation is provided for participation. While individuals may not personally benefit, the study aims to generate feasibility data on voice-based heart rhythm monitoring, potentially reducing reliance on costly consumer devices or frequent clinic visits. Findings will support future large-scale trials and may contribute to improved remote monitoring strategies for atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

To participate in this study, patients must meet all of the following inclusion criteria:

1. Diagnosis of atrial fibrillation and presenting for cardioversion at Allina Health in atrial fibrillation
2. 3. ≥ 18 years of age Written informed consent obtained from patient in English

Exclusion Criteria:

Patients who meet any of the following criteria must be excluded from this study:

1. History of a pacemaker
2. History of dysphasia or difficulty with word finding
3. History of vocal cord dysfunction
4. Patient with atrial flutter as presenting arrhythmia
5. Planned transesophageal echocardiogram (TEE) with cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with a diagnosis of atrial fibrillation scheduled for elective direct-current cardioversion at the Minneapolis Heart Institute Foundation (Abbott Northwestern Hospital). Eligible patients are identified by research staff via EMR pre-screening of cardioversion/procedure and clinic schedules and by provider referral; written informed consent in English is obtained prior to the procedure. Key exclusions: prior pacemaker; dysphasia or word-finding difficulty; vocal cord dysfunction; atrial flutter as the presenting arrhythmia; planned transesophageal echocardiogram (TEE) with cardioversion. No upper age limit. Single-center, single-cohort; no biospecimens collected.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of voice-based rhythm classification vs ECG | Pre-cardioversion (same day), post-cardioversion before discharge (same day), and follow-up at 1 week-1 month post-procedure; overall up to 1 month after cardioversion
  Percentage of Vital Audio (Sauti v1.0) rhythm classifications (regular vs irregular) that match the ECG-determined rhythm at the same time point. Participants serve as their own controls. Results are aggregated across the three time points; 95% confidence intervals will be reported.
Accuracy of voice-based rhythm classification vs ECG | Pre-cardioversion (same day), post-cardioversion before discharge (same day), and follow-up at 1 week-1 month post-procedure; overall up to 1 month after cardioversion
  Percentage of Vital Audio (Sauti v1.0) rhythm classifications (regular vs irregular) that match the ECG-determined rhythm at the same time point. Participants serve as their own controls. Results are aggregated across the three time points; 95% confidence intervals will be reported

IPD SHARING:
Plan to Share IPD: Undecided